CLINICAL TRIAL: NCT01481012
Title: The Epidemiology of Bleeding and Clotting in Patients Undergoing Heart Transplantation, Coronary Artery Bypass Graft Surgery,or Implantation of Left Ventricular Assist Devices
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment - terminated for futility.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-1093 PD; 5P50HL077096 (NIH)
Record Dates: First submitted 2011-11-07; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Congestive Heart Failure
Keywords: Heart transplantation; Coronary artery bypass graft (CABG) surgery; Left ventricular assist device implantation surgeries
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for the following markers of thrombin generation and platelet function will be drawn, spun, aliquoted and stored for later batched analysis: - Thrombo-antithrombin complex (TAT); - Prothrombin Fragment 1+2 (F1.2); - Thromboelastrograph (TEG) (performed at the clinical site when available); - Additional markers of coagulation and platelet activation (for future consideration) - 4ml of plasma frozen in 1ml aliquots.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: Cardiopulmonary Bypass + Heart Transplantation: CPB for orthotopic heart transplantation (excluding any patients with VADs)
- Group II: Cardiopulmonary Bypass + Pulsatile LVAD: CPB for implantation of a Thoratec HeartMate I LVAD (for destination therapy or bridge to transplantation).
- Group III: Cardiopulmonary Bypass + Continuous Flow LVAD: CPB for implantation of an axial flow or centrifugal flow LVAD (for destination therapy or bridge to transplantation) (e.g. HeartMate II, DeBakey VAD or VentraAssist LVAS)
- Group IV: Cardiopulmonary Bypass + CABG Surgery: CPB for CABG surgery

SUMMARY:
The purpose of this study is to obtain data or information on how blood clotting factors are activated during open heart surgery. In particular, the investigators are interested in how blood clotting factors are activated by the heart-lung bypass machine and by left ventricular assist devices (LVAD). Patients on these two machines have an increased risk of bleeding and blood clot formation. This is because both machines stimulate the intrinsic coagulation pathway, one of the chemical pathways that cause blood to clot. The process of surgery itself also stimulates the "extrinsic coagulation pathway," the other chemical pathway that causes blood to clot. Stimulating these coagulation pathways can use up the body's clotting factors. As a result, patients may be at risk for both bleeding and blood clot formation. The investigators would like to study how the blood factors are activated during and after surgery, to help develop treatments to prevent bleeding and clot formation.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study to characterize the epidemiology of bleeding and clotting in patients with underlying systolic ventricular dysfunction undergoing heart transplantation, CABG surgery, or implantation of left ventricular assist devices. Patients will be followed for up to 28 days post-implant, post-CABG, post-heart transplant, or until hospital discharge, whichever comes first. There will be no randomization for this observational study.

We will enroll 100 patients (we expect the distribution to be approximately 30 per Groups I - III, but no cap per group, and 10 for Group IV) who have been scheduled to undergo CPB within 24 hours for one of the following:

Group I: Cardiopulmonary Bypass + Heart Transplantation CPB for orthotopic heart transplantation (excluding any patients with VADs)

Group II: Cardiopulmonary Bypass + Pulsatile LVAD CPB for implantation of a Thoratec HeartMate® I LVAD (for destination therapy or bridge to transplantation)

Group III: Cardiopulmonary Bypass + Continuous Flow LVAD CPB for implantation of an axial flow or centrifugal flow LVAD (for destination therapy or bridge to transplantation) (e.g. HeartMate® II, DeBakey VAD® or VentrAssist® LVAS)

Group IV: Cardiopulmonary Bypass + CABG/Valve Surgery CPB for CABG or valve surgery

Heart transplantation and perioperative care will be performed in accordance with the standard of care at the clinical center. Pulsatile LVAD (e.g. HeartMate® I) implantation and perioperative management will be performed in accordance with the standard of care at the clinical center, and guided by the HeartMate® I Directions for Use. Continuous flow LVAD implantation and perioperative management will be performed in accordance with the standard of care at the clinical center, and guided by the specific VAD manufacturer's Directions for Use. CABG surgery and perioperative care will be performed in accordance with the standard of care at the clinical center.

We anticipate that enrollment will be completed over a six-month period.

We hypothesize that the initial activation of the intrinsic pathway of coagulation is attenuated for several days in patients undergoing CPB for CABG alone; however, in subjects undergoing CPB with VAD implantation or cardiac transplantation, activation of this pathway is biphasic and sustained.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, release of medical information, and HIPAA forms;
2. Age greater than or equal to 18 years;
3. Male, postmenopausal female, or female who may become pregnant but is using adequate contraceptive precautions (defined as oral contraceptive, intrauterine devices, surgical contraception or a combination of a condom and a spermicide), with negative pregnancy test;
4. Admitted to the clinical center at the time of enrollment;
5. Approved and scheduled to undergo one of the following within 24 hours of enrollment:

   * Orthotopic heart transplantation
   * CABG and/or valve surgery on CPB; these patients must have an LV ejection fraction of ≤35%
   * Implantation of a pulsatile LVAD (e.g.Thoratec HeartMate® I LVAD) for destination therapy or bridge to transplantation
   * Implantation of a continuous flow LVAD (e.g. HeartMate® II, DeBakey VAD® or VentrAssist® LVAS) for destination therapy or bridge to transplantation

Exclusion Criteria:

1. History of a platelet disorder;
2. History of a known, or an inherited, or an acquired coagulation disorder in the study subject;
3. Stroke within 30 days prior to enrollment;
4. Allergy to heparin or protamine;
5. Participation in a clinical investigational intervention trial, with the exception of an investigational VAD trial, at the time of enrollment;
6. Received investigational intervention within 30 days of enrollment, with the exception of an investigational VAD trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with underlying systolic ventricular dysfunction who will undergo heart transplantation, CABG surgery, implantation of a pulsatile LVAD, or implantation of a continuous flow LVAD (as destination therapy or bridge to transplantation) within 24 hours of enrollment, are candidates for this study.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Thrombin Generation Markers | At time of surgery (before initiation of Cardiopulmonary Bypass)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | At time of surgery (dismantling the sterile environment)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 1
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | At time of surgery
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day12 (while remaining in hosp)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 16 (while remaining in hosp)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 20 (while remaining in hosp)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 24 (while remaining in hosp)
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.

SECONDARY OUTCOMES:
Bleeding | At time of surgery (dismantling of the sterile environment)
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 1
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 12 (± 3 days) (or at time of discharge, whichever comes first)
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 20 (± 3 days) (or at time of discharge, whichever comes first)
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 28 (± 3 days) (or at time of discharge, whichever comes first)
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Coagulation Markers | At time of surgery ( before initiation of Cardiopulmonary Bypass)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | At time of surgery (dismantling the sterile environment)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 1
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | At time of surgery
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 12 (while remaining in hosp)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 16 (while remaining in hosp)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 20 (while remaining in hosp)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 24 (while remaining in hosp)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 28 (± 3 days) (or at time of discharge, whichever comes first)
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Serious Adverse Events | Duration of the Study, up to 28 days post-implant, post-CABG, post heart-transplant, or until hospital discharge, whichever comes first.
  The incidence and frequency of all expected and unexpected serious adverse events will be determined. Since this is an observational study, there will be no adverse events directly attributable to a study intervention. However, adverse events that may potentially contribute to the risk or course of bleeding and clotting in patients undergoing heart transplantation, CABG surgery, or implantation of LVADs will be monitored. The adverse events are defined according to the definitions recently finalized by the INTERMACS LVAD registry.
Thrombin Generation Markers | Post-operative day 2
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 3
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 4
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombo Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 5
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombo Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 6
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Thrombin Generation Markers | Post-operative day 7
  We will compare the following endpoints among the cardiac transplant, CABG, and LVAD recipients:
  Thrombin Generation Markers: Assays will be performed to quantify the levels of the following markers at the specified time points: Thrombo-antithrombin complex (TAT), Prothrombin Fragment 1 +2 (F1.2), and Thromboelastography (TEG) will be performed when available to assess platelet function.
Bleeding | Post-operative day 2
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 3
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 4
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 5
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 6
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Bleeding | Post-operative day 7
  Bleeding will be assessed by measurement of units of packed red blood cells (or whole blood) transfused from initiation of the procedure through the 24 hour post-operative period following LVAD implantation, heart transplantation, or CABG. In addition, we will measure transfusion requirements through the 28 day post-operative period. Units of additional blood products transfused will also be measured, including FFP, cryoprecipitate, and platelets. Hemoglobin, hematocrit and platelet count will be measured as an indirect assessment of blood loss.
Coagulation Markers | Post-operative day 2
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 3
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 4
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 5
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 6
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.
Coagulation Markers | Post-operative day 7
  Assays will be performed to assess the levels of following coagulation markers: Prothrombin time (PT) with (INR), Partial thromboplastin time (PTT), Complete Blood Count (CBC) including hemoglobin, hematocrit, and platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Desvigne-Nickens, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Yoshifumi Naka, MD, Study Chair — Columbia University; Annetine Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sharp Memorial Hospital, San Diego, California
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia Presbyterian Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - LDS Hospital, Salt Lake City, Utah
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin